CLINICAL TRIAL: NCT00929773
Title: Study of the Effect of Low Level Laser Light Therapy on the Reduction of Chronic Pain of the Neck and Shoulders
Brief Title: Low Level Laser Therapy to Reduce Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECP-001
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia PL2000 Laser (Active Comparator): Low level laser light energy comprised of 1 milliWatts (mW) of red light (635 nm).
  Interventions: Device: Erchonia PL2000 Laser
- Placebo laser (Placebo Comparator): inactive light
  Interventions: Device: Placebo laser

INTERVENTIONS:
Device: Erchonia PL2000 Laser — Low level laser light therapy device that emits 1 mW of red (635 nm wavelength) light. It is a hand-held device that uses rechargeable batteries or a separate power adapter.
  Other Names: Erchonia PL5000; Erchonia EVRL Laser
  Arms: Erchonia PL2000 Laser
Device: Placebo laser — Inactive laser light.
  Arms: Placebo laser

SUMMARY:
The purpose of this study was to determine whether low level laser light directed at the neck and shoulders could be effective in the temporary reduction of chronic pain in the neck and shoulder region.

DETAILED DESCRIPTION:
Chronic neck and shoulder pain arising from osteoarthritis, chronic muscle spasms or thoracic or cervical spine sprain strain can be seriously debilitating. Currently available treatment options such as pain relief medication, ice pack, massage, physical therapy and chiropractic are typically of limited effectiveness. More permanent options such as surgery are invasive with long recovery periods and side-effects and complications of their own. Low level laser light therapy, with its proven anti-inflammatory ability, offers a simple non-invasive option for the reduction of chronic neck and shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Muscular-skeletal pain in the neck/shoulder region
* Acute and chronic pain in the neck/shoulder region
* Restricted range of motion in the neck/shoulder region
* Fibrosis or scar tissue in the neck/shoulder region
* Inflammation in the neck/shoulder region
* Altered function in the neck/shoulder region
* Muscle strains in the neck/shoulder region
* Rating of 30 or greater on the 0-100 Visual Analog Scale (VAS) pain scale
* 18-65 years of age

Exclusion Criteria:

* Severely herniated disks
* Pregnancy
* Taken pain medication within the past 12 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-07; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Amy, DC, Principal Investigator; George Gonzalez, DC, Principal Investigator; John Pinto, DC, Principal Investigator; Allen Wentworth, DC, Principal Investigator; Robert Stashko, DC, Principal Investigator

REFERENCES:
- See also: FDA 510(k)#K050672 clearance listing for pain reduction — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=17825
- See also: FDA 510(k)#K012580 clearance based on these study results — http://www.accessdata.fda.gov/cdrh_docs/pdf/K012580.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was July through September, 2000 at a single medical clinic.
Pre-assignment Details: Following enrollment and prior to group assignment, study participants underwent study qualification evaluation which included a self-report rating of current neck and/or shoulder pain level on the 0-100 VAS.
Groups:
- Erchonia PL2000 Laser: Low level laser energy comprised of 1 milliWatt (mW) of near-infrared light (635 nm) to the neck and shoulder area .
Period: Overall Study
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erchonia Low Level Laser Therapy: Low level laser energy comprised of 1 mw of near-infrared light (635 nm) to the neck and shoulder area .
- Total: Total of all reporting groups
Arm/Group | Erchonia Low Level Laser Therapy | Placebo Laser | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 25 | 25 | 50
Location of Pain [Number; unit: participants] — Subject report of pain located in the neck, shoulder or both regions.
  participants
    Shoulders | 10 | 14 | 24
    Neck | 13 | 14 | 27
    Neck & Shoulders | 27 | 22 | 49
Type of Pain [Number; unit: participants]
  Chronic | 43 | 44 | 87
  Acute | 7 | 6 | 13
Pain Rating on the Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Scale (VAS) is used as a self-reported measure of current pain level. Participants mark the spot on the line scale that shows the level of their pain at that time. The scale ranges fron '0: no pain at all' to '100: worst pain imaginable.' The scale is a straight line of 100mm. The point marked by the participant is measured as their current pain level. The higher the number, the greater the pain level. To qualify to be in the study, participants needed to record a Baseline pain level on the VAS of 30 or greater.
  units on a scale | 51.14 (16.50) | 49.06 (19.48) | 50.10 (18.00)
Duration of Pain [Mean (Standard Deviation); unit: months] | 57.11 (121.40) | 40.25 (71.13) | 48.15 (97.64)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Self-reported Degree of Pain on the Visual Analog Scale (VAS) in the Neck and Shoulder Area Decreased by 30% or More From Before to After Study Treatment.
Description: Self-reported degree of pain in the neck and shoulder region on the Visual Analog Scale (VAS). The VAS is a 100 mm long horizontal line ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. Participants mark a point along the line that best represents the pain they are experiencing at that moment.
Time Frame: baseline and one hour
Measure: Number; unit: participants
Groups:
- Erchonia PL2000 Laser: Low level laser energy comprised of 1 mW of near-infrared light (635 nm) to the neck and shoulder area .
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
participants | 40 | 7
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Change in Range of Motion (ROM) for the Left Side of the Neck From Baseline to One Hour After Study Treatment.
Description: Range of motion (ROM) for the left side of the neck is a measure of how well the neck can move to the left side. The participant gently tilts their neck to the left side as far as possible, and this distance is measured in degrees. The change for ROM for the left side of the neck is measured as the difference in degrees of ROM recorded from baseline to one hour after study treatment. If the change is positive (+), this means that ROM has gotten better and the neck can move further to the left side than before getting the treatment. If the change is negative (-), this means that ROM has gotten worse and the neck can move less to the left side than before getting the treatment
Time Frame: baseline and one hour
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Erchonia PL2000 Laser: Low level laser energy comprised of 1 mW of near-infrared light (635 nm) to the neck and shoulder area.
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
degrees | 11.28 (9.64) | 0.02 (6.90)
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < .0001, t-test, 2 sided

3. Secondary Outcome: Change in Range of Motion (ROM) for the Left Shoulder From Baseline to One Hour After Study Treatment.
Description: Range of motion (ROM) for the left shoulder is a measure of how well the participant can move the left shoulder. The participant gently raises the left shoulder (and left arm) as far as possible, and this distance is measured in degrees. The change for ROM for the left shoulder is measured as the difference in degrees of ROM recorded from baseline to one hour after study treatment. If the change is positive (+), this means that ROM has gotten better and can move the left shoulder better and further than before getting the treatment. If the change is negative (-), this means that ROM has gotten worse and the left shoulder can move less easily and not as far than before getting the treatment
Time Frame: one hour
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
degrees | 28.00 (22.67) | 2.24 (0.33)
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Primary Outcome: Change in Self-reported Degree of Pain in the Neck-shoulder Region on the 0-100 Visual Analog Scale (VAS)
Description: Self-reported degree of pain in the neck and shoulder region on the Visual Analog Scale (VAS). The VAS is a 100 mm long horizontal line ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. Participants mark a point along the line that best represents the pain they are experiencing at that moment. The change is calculated as the difference from the VAS score recorded at baseline to the VAS score recorded one hour after study treatment administration. A positive change (+) means that the pain got worse and a negative change (-) means that the pain got better.
Time Frame: baseline and one hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
units on a scale | -27.38 (19.28) | -2.43 (12.57)
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Change in Range of Motion (ROM) for the Right Side of the Neck From Baseline to One Hour After Study Treatment.
Description: Range of motion (ROM) for the right side of the neck is a measure of how well the neck can move to the right side. The participant gently tilts their neck to the right side as far as possible, and this distance is measured in degrees. The change for ROM for the right side of the neck is measured as the difference in degrees of ROM recorded from baseline to one hour after study treatment. If the change is positive (+), this means that ROM has gotten better and the neck can move further to the right side than before getting the treatment. If the change is negative (-), this means that ROM has gotten worse and the neck can move less to the right side than before getting the treatment.
Time Frame: baseline and one hour
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
degrees | 11.06 (9.63) | 0.72 (7.58)
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Change in Range of Motion (ROM) for the Right Shoulder From Baseline to One Hour After Study Treatment.
Description: Range of motion (ROM) for the right shoulder is a measure of how well the participant can move the right shoulder. The participant gently raises the right shoulder (with right arm) as far as possible, and this distance is measured in degrees. The change for ROM for the right shoulder is measured as the difference in degrees of ROM recorded from baseline to one hour after study treatment. If the change is positive (+), this means that ROM has gotten better and the right shoulder can move further more easily than before getting the treatment. If the change is negative (-), this means that ROM has gotten worse and the right shoulder can move less and not as far to the left side than before getting the treatment.
Time Frame: baseline and one hour
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Erchonia PL2000 Laser | Placebo Laser
Number analyzed (Participants) | 50 | 50
degrees | 30.90 (25.97) | 1.70 (11.60)
Statistical Analysis 1: Comparison: Erchonia PL2000 Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Erchonia Low Level Laser Therapy | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No